CLINICAL TRIAL: NCT05905237
Title: Effects of Laser Species and Ocular Antioxidant Activity on Postoperative Inflammation and Visual Prognosis in Patients Undergoing Ophthalmic Surgery - a Comparative Study
Brief Title: Measurement of Antioxidant Activity on Postoperative Inflammation in Patients Undergoing Ophthalmic Surgery
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Nobel Eye Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202200858B0A3
Record Dates: First submitted 2023-05-26; First posted 2023-06-15 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2023-07

CONDITIONS: Cataract; Myopia
Keywords: antioxidants
MeSH Terms: conditions — Cataract; Myopia | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tears are collected using Schirmer Tear Test Strips before and after surgery. Patients undergoing intraocular surgery lose their aqueous humor due to full thickness wounds. During operation, approximately 0.1-0.5 mL of the humor is collected into a microcentrifuge tube, and then, the humor leaked from wound at one day after surgery is also collected with an ophthalmic sponge. During the SMILE procedure, a sample of the corneal len (lenticule) will be produced, which is also placed in a microcentrifuge tube. All the above specimens were temporarily stored in liquid nitrogen and sent to the laboratory of the Research Building of Linkou Chang Gung Hospital on the day of acquisition for storage in a -80℃ refrigerator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Cataract surgery, Femtosecond-LASIK, SMILE — Cataract surgery includes both conventional and femtosecond laser assisted. Femtosecond-LASIK and SMILE are options for patients to correct myopia.

SUMMARY:
This trial hypothesized that novel laser refractive surgery techniques (PRK, LASIK, SMILE) or laser-assisted cataract surgery (FLACAS) could suppress postoperative inflammation and improve recovery in patients by reducing oxidative stress generated by the surgical procedure. It is also intended to verify whether the new laser technology is necessary for clinical use in groups with low antioxidant activity through the detection of antioxidant activity in the eyes of patients.

ELIGIBILITY:
Inclusion Criteria:

* over 20 years old (included)
* corneal refractive surgery or cataract surgery patients

Exclusion Criteria:

* patients with eye infections
* presence of severe retinal disease
* presence of severe eye injury or severe ptosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A prospective, non-randomized trial was conducted at the Nobel Eye Clinic. This study included patients with the following conditions: (1) older than 20 years old (inclusive), (2) expected to undergo corneal refractive surgery or cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Change of Total Antioxidant Capacity (TAC) in tears from Baseline to 1 week after surgery. | Before the operation and 1 week after surgery.
Change of Total Antioxidant Capacity (TAC) in tears from Baseline to 1 month after surgery. | Before the operation and 1 month after surgery.
Change of Total Antioxidant Capacity (TAC) in tears from Baseline to 3 months after surgery. | Before the operation and 3 months after surgery.
Change of Total Antioxidant Capacity (TAC) in tears from Baseline to 6 months after surgery. | Before the operation and 6 months after surgery.
Change of Ascorbic Acid (AA) in tears from Baseline to 1 week after surgery. | Before the operation and 1 week after surgery.
Change of Ascorbic Acid (AA) in tears from Baseline to 1 month after surgery. | Before the operation and 1 month after surgery.
Change of Ascorbic Acid (AA) in tears from Baseline to 3 months after surgery. | Before the operation and 3 months after surgery.
Change of Ascorbic Acid (AA) in tears from Baseline to 6 months after surgery. | Before the operation and 6 months after surgery.
Change of Total Antioxidant Capacity (TAC) in aqueous humor from Baseline to one day after surgery. | During the operation and one day after surgery.
Change of Ascorbic Acid (AA) in aqueous humor from Baseline to one day after surgery. | During the operation and one day after surgery.

SECONDARY OUTCOMES:
Examination of best corrected visual acuity (BCVA). | Before the operation.
Examination of uncorrected visual acuity (UCVA). | Before the operation.
Examination of uncorrected visual acuity (UCVA). | One week after surgery.
Examination of uncorrected visual acuity (UCVA). | One month after surgery.
Examination of intraocular pressure (IOP). | Before the operation.
Examination of intraocular pressure (IOP). | One week after surgery.
Examination of intraocular pressure (IOP). | One month after surgery.
Examination of central corneal thickness (CCT). | Before the operation.
Examination of central corneal thickness (CCT). | One week after surgery.
Examination of central corneal thickness (CCT). | One month after surgery.
Examination of axial length (AXL). | Before the operation.
Examination of anterior chamber depth (ACD). | Before the operation.
Examination of lens thickness (LT). | Before the operation.
Examination of manifest refraction. | Before the operation.
Examination of manifest refraction. | One week after surgery.
Examination of manifest refraction. | One month after surgery.
Examination of corneal curvature. | Before the operation.
Examination of corneal curvature. | One week after surgery.
Examination of corneal curvature. | One month after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Chi Chen, PhD, Study Chair — Chang Gung Memorial Hospital
Locations (2):
- Taiwan (2):
  - ChangGungMH, Taoyuan District, Taoyuan City
  - Nobel Eye Institute, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barati E, Nikzad H, Karimian M. Oxidative stress and male infertility: current knowledge of pathophysiology and role of antioxidant therapy in disease management. Cell Mol Life Sci. 2020 Jan;77(1):93-113. doi: 10.1007/s00018-019-03253-8. Epub 2019 Aug 3. PMID 31377843
- [Background] Sacca SC, Roszkowska AM, Izzotti A. Environmental light and endogenous antioxidants as the main determinants of non-cancer ocular diseases. Mutat Res. 2013 Apr-Jun;752(2):153-171. doi: 10.1016/j.mrrev.2013.01.001. Epub 2013 Jan 19. PMID 23337404
- [Background] Moreau KL, King JA. Protein misfolding and aggregation in cataract disease and prospects for prevention. Trends Mol Med. 2012 May;18(5):273-82. doi: 10.1016/j.molmed.2012.03.005. Epub 2012 Apr 19. PMID 22520268
- [Background] Spector A. Review: Oxidative stress and disease. J Ocul Pharmacol Ther. 2000 Apr;16(2):193-201. doi: 10.1089/jop.2000.16.193. PMID 10803430
- [Background] Rosado-Adames N, Afshari NA. The changing fate of the corneal endothelium in cataract surgery. Curr Opin Ophthalmol. 2012 Jan;23(1):3-6. doi: 10.1097/ICU.0b013e32834e4b5f. PMID 22134364
- [Background] Kim EC, Meng H, Jun AS. N-Acetylcysteine increases corneal endothelial cell survival in a mouse model of Fuchs endothelial corneal dystrophy. Exp Eye Res. 2014 Oct;127:20-5. doi: 10.1016/j.exer.2014.06.002. Epub 2014 Jun 18. PMID 24952277
- [Background] Kimoto M, Shima N, Yamaguchi M, Amano S, Yamagami S. Role of hepatocyte growth factor in promoting the growth of human corneal endothelial cells stimulated by L-ascorbic acid 2-phosphate. Invest Ophthalmol Vis Sci. 2012 Nov 9;53(12):7583-9. doi: 10.1167/iovs.12-10146. PMID 23081981
- [Background] M Padua IR, P Valdetaro G, B Lima T, K Kobashigawa K, E S Silva P, Aldrovani M, M Padua PP, Laus JL. Effects of intracameral ascorbic acid on the corneal endothelium of dogs undergoing phacoemulsification. Vet Ophthalmol. 2018 Mar;21(2):151-159. doi: 10.1111/vop.12490. Epub 2017 Jul 17. PMID 28714237
- [Background] Hsueh YJ, Meir YJ, Yeh LK, Wang TK, Huang CC, Lu TT, Cheng CM, Wu WC, Chen HC. Topical Ascorbic Acid Ameliorates Oxidative Stress-Induced Corneal Endothelial Damage via Suppression of Apoptosis and Autophagic Flux Blockage. Cells. 2020 Apr 11;9(4):943. doi: 10.3390/cells9040943. PMID 32290365
- [Background] Horwath-Winter J, Kirchengast S, Meinitzer A, Wachswender C, Faschinger C, Schmut O. Determination of uric acid concentrations in human tear fluid, aqueous humour and serum. Acta Ophthalmol. 2009 Mar;87(2):188-92. doi: 10.1111/j.1755-3768.2008.01215.x. Epub 2008 Jun 11. PMID 18547277
- [Derived] Chen HC, Yang SF, Lee CY, Hsueh YJ, Huang JY, Chang CK. Differences in change of post-operative antioxidant levels between laser-assisted lenticule extraction and femtosecond laser in situ keratomileusis. J Cell Mol Med. 2024 Jan;28(2):e18069. doi: 10.1111/jcmm.18069. Epub 2023 Dec 5. PMID 38051678